CLINICAL TRIAL: NCT03481166
Title: Empowering Women to Cope with Breastfeeding Pain: a Feasibility Randomized Controlled Trial of an Educational Anticipatory Guidance Intervention
Brief Title: Women Empowered Through Education to Breastfeed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Women's College Hospital (Other)
Responsible Party: Principal Investigator, Kim Jackson, Assistant Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 111412
Record Dates: First submitted 2018-02-14; First posted 2018-03-29 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Breastfeeding; Pain; Nipple Pain During Lactation
Keywords: pilot; randomized controlled trial; prenatal education; anticipatory guidance
MeSH Terms: conditions — Breast Feeding; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Education on breastfeeding pain (Experimental): Both the experimental and control groups will receive usual prenatal education offered through our regional public health program. In addition to usual prenatal education, the experimental group will also receive a one-hour, nurse led (a Registered Nurse specially trained in perinatal care), small group-based education session with specific focus on breastfeeding pain. The goals of this educational intervention are to provide pregnant women with anticipatory guidance around pain which is commonly experienced while breastfeeding in the first two weeks postpartum. Education will include the prevalence, etiology and management of various types of breastfeeding-related pain experienced postpartum.
  Interventions: Other: Education on breastfeeding pain
- Usual prenatal education (No Intervention): Women allocated to the usual prenatal education group will receive prenatal classes through their local public health unit. Women enrolled in classes will receive approximately 12 hours of combined in-class and online prenatal content. Topics include: discomforts of pregnancy, labor and birth, medical interventions, adjustment to parenting, breastfeeding, and caring for the newborn. Breastfeeding-related material includes basic mechanisms of milk production, benefits of breastfeeding, benefits of skin-to-skin, correct breastfeeding latch, breastfeeding positions, timing of feeds, responding to infant cues, and caring for nipples. Women in the usual prenatal education group will not receive education on the prevalence and etiology of nipple pain, nor specific pain management strategies.

INTERVENTIONS:
Other: Education on breastfeeding pain — A Registered Nurse with specialization in antenatal and postpartum care will deliver a one-hour, group-based educational session specifically on breastfeeding-related pain, including: common causes of nipple pain, prevalence of nipple pain, impact of pain on milk ejection reflex, and common approaches to prevention and management of nipple pain.
  Arms: Education on breastfeeding pain

SUMMARY:
The experience of breastfeeding-related pain is common for postpartum women, but is not often anticipated as part of the postpartum experience. This feasibility randomized controlled trial aims to examine the effectiveness of a nurse-led educational intervention using anticipatory guidance among pregnant women wishing to breastfeed on breastfeeding outcomes, breastfeeding-related pain, and maternal satisfaction.

DETAILED DESCRIPTION:
Despite the relative ubiquity of breastfeeding-related pain, exploratory studies suggest women are largely unprepared for breastfeeding-related pain in the early postpartum period [1-3]. In turn, postpartum women often experience an incongruence between how breastfeeding is idealized by Western society, and the reality of their early breastfeeding experiences. Furthermore, painful breastfeeding experiences serve to intensify this incongruity and may lead to disillusionment, feelings of negative self-worth and premature breastfeeding cessation [1,3]. As such, the overarching goals of this one-year project are to compare usual prenatal education to anticipatory guidance to: 1) examine the effectiveness of a breastfeeding education session using anticipatory guidance on breastfeeding outcomes and satisfaction during the postpartum period; and 2) test the feasibility of the methods and procedures needed for the successful implementation and validity of a full-scale randomized controlled trial (RCT). This one-year project has 5 objectives:

To fill a knowledge gap in nursing and allied health-related literature by examining the effect of a one-hour, nurse-led, breastfeeding education session using anticipatory guidance during pregnancy on: Objective 1: breastfeeding duration and exclusivity versus those receiving usual prenatal education; Objective 2: overall satisfaction with the educational experience versus those receiving usual prenatal education; Objective 3: breastfeeding self-efficacy and infant feeding attitudes; Objective 4: postpartum breastfeeding-related pain and; Objective 5: To determine if this intervention study protocol is practical (e.g., accrual rates, satisfaction, compliance, sample size) and to test the process, resources, management and scientific basis [4] for a future, full-scale RCT.

Forty pregnant women enrolled in prenatal classes provided by the Middlesex London Health Unit (MLHU) and who are intending to breastfeed will be enrolled in this feasibility randomized controlled trial.

Following ethics approval, interested pregnant women who have enrolled in/awaiting antenatal classes at the MLHU will contact the RA to discuss the study. Interested women will be screened for eligibility, and if eligible and consenting, baseline data will be collected. Participants will then be randomized to either intervention (n=20) or control group (n=20). Randomization will be achieved by using sealed, opaque, sequentially numbered envelopes containing randomly generated numbers, prepared by an RA external to the study. An RA will open the next sequentially numbered envelope and reveal the group allocation to the participant. The control group will receive usual antenatal education provided to all women who enroll in MLHU prenatal classes. The intervention group will receive an additional one-hour 'booster session' (by a perinatal RN) of antenatal education specifically focused on the postpartum experience of breastfeeding, including anticipatory guidance around breastfeeding-related pain, and management strategies. To control for contamination, women who have peers/family already in the study will be excluded. An emailed link to a follow-up questionnaire will be sent at 2 and 4 weeks postpartum to determine if they are breastfeeding or not, breastfeeding exclusivity, level of breastfeeding-related pain, breastfeeding self-efficacy, maternal attitudes toward infant feeding, and maternal satisfaction with antenatal education.

ELIGIBILITY:
Inclusion Criteria:

Women who self-enrolled in prenatal education classes at public health unit who:

* Can read and write in English
* Less than or equal to 32 weeks gestation (in pregnancy)
* Planning to breastfeed their infant
* 19 years of age or older
* Internet accessible

Exclusion Criteria:

* Greater than 32 weeks gestation
* have been identified as having a high-risk pregnancy
* have self-identified barriers to breastfeeding
* have peers or family already enrolled in the study

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Breastfeeding duration | 4 weeks postpartum
  Breastfeeding duration will be measured by asking women if they have breastfed in the past 24 hours or not. If a participant has stopped breastfeeding, they will be asked for the last date they breastfed their infant to determine the number of days (duration) of breastfeeding.

SECONDARY OUTCOMES:
Breastfeeding exclusivity | 2 and 4 weeks postpartum
  Breastfeeding exclusivity is defined as the receipt of breast milk only with no additional food or liquid, including water. Breastfeeding exclusivity will be categorized according to the World Health Organization Infant and Young Child Feeding guidelines (2009) with the following categories: exclusive breastfeeding, predominant, complimentary feeding, breastfeeding or bottle-feeding. Among the extant breastfeeding literature, this is the most commonly utilized means to measure breastfeeding exclusivity.
Pain severity | 4 weeks postpartum
  Pain severity will be measured using an 11-point numeric rating scale, where zero represents no pain, and 10 represents the worst pain imaginable.

OTHER OUTCOMES:
maternal satisfaction | 2 and 4 weeks postpartum
  Women's self-report of satisfaction with the education they received will be measured by asking women: "were you satisfied receiving additional breastfeeding education", "how effective was the breastfeeding education session in helping you to breastfeed your baby", "how effective was the additional breastfeeding education session in helping you to anticipate the possibility of breastfeeding pain". Responses will include descriptions on a 5 point Likert scale. For example, "1" for "very satisfied", and "5 for "very dissatisfied". There are no reliable, validated measurement tools measuring maternal satisfaction in this context.
breastfeeding self-efficacy | 2 and 4 weeks postpartum
  Self reported maternal breastfeeding self-efficacy will be measured using the Breastfeeding self-efficacy scale short form (Dennis, 2003. The breastfeeding self-efficacy scale: psychometric assessment of the short form. J Obstet Gynecol Neonatal Nurs, 32(6), 734-44)
women's attitude toward breastfeeding | 2 and 4 weeks postpartum
  Self reported maternal attitude toward breastfeeding will be measured using the Iowa Infant Feeding Attitude Scale (De la Mora et al., 1999. The Iowa Infant Feeding Attitude Scale: Analysis of reliability and validity. Journal of Applied Social Psychology, 29(11), 2362-2380)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley T Jackson, PhD, Principal Investigator — Western University
Locations (1):
- Middlesex London Health Unit, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No